CLINICAL TRIAL: NCT06759012
Title: Study on the Medical Education Capability of the EyeTeacher Artificial Intelligence Platform
Acronym: EyeTeacher
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: THU01-20240100
Record Dates: First submitted 2024-12-05; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Medical Education
Keywords: Medical education; Multimodality AI; Generative AI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Attend EyeTeacher lecture before taking the regular ophthalmology lecture in medical school.
  Interventions: Other: EyeTeacher
- Control group (No Intervention): Attend regular ophthalmology lectures in medical school.

INTERVENTIONS:
Other: EyeTeacher — Participants randomized to the intervention group will receive access to the EyeTeacher system, along with their username, password, and a user manual, one week before the start of the course. They will follow instructions on the website and complete a quiz before and after each course. After completing the EyeTeacher curriculum, they will take the first examination (Examination 1) and complete a set of questionnaires. A classroom will be provided for study purposes, but no restrictions will be imposed on the study location. Following the EyeTeacher section, participants will attend the ophthalmology course in the regular training program, with support from the EyeTeacher system. They will be evaluated according to the ophthalmology posting's evaluation criteria (Examination 2).
  Arms: Interventional group

SUMMARY:
With the rise of generative artificial intelligence and large language models, medical education is undergoing a significant transformation. Numerous studies have highlighted the limitations of traditional educational knowledge acquisition and the potential impact of artificial intelligence on medical education, resident training, and continuing education for clinical practitioners. However, there is a lack of real-world experiments on the effectiveness of AI-integrated education.

Artificial intelligence can provide extensive educational resources and tools that are not limited by geographical location or language, thereby lowering the barrier to accessing high-quality medical education and promoting educational equity. Nevertheless, the performance of AI models trained by different medical institutions or healthcare systems may vary.

To offer a more universal, accessible, high-quality, and interconnected educational journey. We have developed a virtual ophthalmology teacher, which developed based on foundational model and large language models. This model, named EyeTeacher provide comprehensive theoretical knowledge and clinical skills enhancement for untrained medical students. To verify the effectiveness of our EyeTeacher across different national ophthalmology education systems and languages, we plan to implement a randomized controlled trial. This trial will assess the clinical capabilities of all participants and explore the advantages and disadvantages of the system compared to traditional teaching methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical medical students who have not taken ophthalmology courses
* Age 21-40
* Gender not restricted
* Sign the informed consent form

Exclusion Criteria:

* Refusal of the research protocol.
* Participants unwilling or unable to understand and complete the questionnaire.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Grade of ophthalmology examination | 1 day after complete lectures
  Title: Ophthalmology Theoretical Examination. The examination includes 40 multiple-choice questions and two essay questions related to ophthalmology knowledge, to be completed within one hour without the use of reference materials. The exam will be graded by experts based on a standardized answer key. The score ranges from 0 to 100, with a higher score indicating a deeper understanding of the ophthalmology knowledge.
  Students in both the interventional group and the control group will complete the exam within the specified time on the EyeTeacher system. The data will be collected in the system's backend.

SECONDARY OUTCOMES:
Time of studying ophthalmology | 1 day after complete lectures
  The study time spent using each teaching module in the interventional group is tracked by the EyeTeacher system website, while the study time for the control group and the out-of-system study time for the interventional group are collected through a questionnaire.
  Questionnaire title: Time of Study in Ophthalmology The questionnaire consists of fill-in-the-blank questions, with time measured in minutes. The content includes: class time, exercise time, discussion time, and reading reference material time. The questionnaires for both the interventional and control groups are completed on the EyeTeacher system, and the data is collected through the backend.
Feedback of teaching from students | 1 day after complete lectures
  Questionnaire title: Feedback of Study in Ophthalmology:
  The Likert scale is used for scoring. The topics include students' evaluations of course design, teacher guidance, empathy, as well as students' self-assessment and evaluation of their interest in ophthalmology.
  The questionnaires for both the interventional and control groups are completed on the EyeTeacher system, and the data is collected through the backend.

CONTACTS AND LOCATIONS:
Locations (7):
- University of Melbourne, Melbourne, Victoria, Australia
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China
- University of Ghana, Accra, Greater Accra Region, Ghana
- Sankara Nethralaya, Chennai, Tamil Nadu, India
- University of Malaya, Kuala Lumpur, Malaysia
- Duke-NUS medical school, Singapore, Singapore
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He B, Kwan AC, Cho JH, Yuan N, Pollick C, Shiota T, Ebinger J, Bello NA, Wei J, Josan K, Duffy G, Jujjavarapu M, Siegel R, Cheng S, Zou JY, Ouyang D. Blinded, randomized trial of sonographer versus AI cardiac function assessment. Nature. 2023 Apr;616(7957):520-524. doi: 10.1038/s41586-023-05947-3. Epub 2023 Apr 5. PMID 37020027
- [Background] Benitez TM, Xu Y, Boudreau JD, Kow AWC, Bello F, Van Phuoc L, Wang X, Sun X, Leung GK, Lan Y, Wang Y, Cheng D, Tham YC, Wong TY, Chung KC. Harnessing the potential of large language models in medical education: promise and pitfalls. J Am Med Inform Assoc. 2024 Feb 16;31(3):776-783. doi: 10.1093/jamia/ocad252. PMID 38269644